CLINICAL TRIAL: NCT03190109
Title: Analyses of Bone Age Determined by Ultrasound in a Cohort of Brazilian Control Children and Adolescents: Comparison With Conventional Bone Age Determined by X-Ray
Brief Title: Bone Age Determined by Ultrasound (BAUS) in Brazilian Control Children
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Faculdade de Ciências Médicas da Santa Casa de São Paulo (Other)
Responsible Party: Principal Investigator, Carlos Alberto Longui, Full Professor, Faculdade de Ciências Médicas da Santa Casa de São Paulo
Other Study IDs: 53659316.3.0000.5479
Record Dates: First submitted 2017-06-12; First posted 2017-06-16 (Actual); Last update posted 2017-06-16 (Actual); Status verified 2017-06

CONDITIONS: Control, Population
Keywords: bone age measurement; skeletal age measurement; ultrasound; x-Ray

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Aiming to validate the use of bone age determined by ultrasound (BAUS) in Brazilian children, normal control students will be studied. X-Ray bone age (RXBA) and BAUS will be determined in 500 children and adolescents of both genders, with chronological age varying from 6-16 years.

Concordance analysis and the correlation between both BA determination methods will be performed.

DETAILED DESCRIPTION:
Bone age is a valuable method to recognize the maturation status of development and growth. Classical analyses is performed by using the Greulich and Pyle X-Ray measurement. Such analyses have some restrictions such as intra- and inter observer variability, and variable synchronicity of bone maturation.

Bone age determined by ultrasound (BAUS) has been indicated as a fast and reproducible method, allowing decimal BA determination and avoiding the need for X-Ray.

Our aim is to validate the BAUS method in Brazilian normal controls. School students of both genders, with age varying from 6 to 16 years will be included.

ELIGIBILITY:
Inclusion Criteria:

* absence of chronic illness and drug ingestion

Exclusion Criteria:

* any chronic disease or medicine use
* body mass index: < -2SDS or > +2SDS
* stature : < -2SDS or > +2SDS

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: normal control school students
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2016-10-13 (Actual); Primary Completion 2017-09 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
bone age determination by ultrasound (BAUS) | chronological ages between 6 and 16 years of age
  Determination of bone age in years by employing a ultrasound device

CONTACTS AND LOCATIONS:
Overall Officials: Carlos A Longui, MD; PhD, Principal Investigator — Full Professor. Head of Pediatric Endocrinology Unit
Locations (1):
- Santa Casa SP - School of Medical Sciences, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No